CLINICAL TRIAL: NCT00331188
Title: The Early Use of Sanvar® With Endoscopic Treatment for the Control of Acute Variceal Bleeding Due to Portal Hypertension
Brief Title: Use of Sanvar® With Endoscopic Treatment for the Control of Acute Variceal Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiovision (Industry)
Responsible Party: Marco Petrella, M.Sc., Ph.D. - Director, Clinical Affairs & New Product Development, Debiovision
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEBV-VAP/EVB-301
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Esophageal Varices; Portal Hypertension; Gastric Varices; Esophageal Bleeding
Keywords: Esophageal Variceal Bleeding; Portal Hypertension; Hepatic Cirrhosis; Cirrhosis; Liver Cirrhosis; Somatostatin Analog; Vapreotide; Acute Esophageal Variceal Bleeding
MeSH Terms: conditions — Esophageal and Gastric Varices; Hypertension, Portal; Liver Cirrhosis; Fibrosis | interventions — vapreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sanvar® (vapreotide)

SUMMARY:
The main objective of this study is to determine the efficacy of early administration of Sanvar® in combination with endoscopic treatment for the control of acute variceal bleeding.

DETAILED DESCRIPTION:
This is a single-arm open-label clinical study with historical controls using Sanvar® (vapreotide) administered for 5 days in patients with acute variceal bleeding due to portal hypertension.

Cirrhotic patients with a history of acute hematemesis and/or melena admitted to the emergency unit and meeting the eligibility criteria will receive, as soon as possible after admission (within a maximum of 24 hours after onset of hemorrhage and within 6 hours after admission), Sanvar® (vapreotide acetate) 50 µg IV bolus followed by an IV continuous infusion of 50 µg/h for 5 days.

The diagnostic and therapeutic endoscopy will be performed as soon as possible after the initiation of the study drug infusion, but no more than 12 hours after the patient's admission to the study center. A final follow up will be performed on Day 42.

Patients for whom the source of bleeding is determined at endoscopy to be due to a cause other than portal hypertension (e.g. gastric ulcer) will be replaced. In addition, in such cases the study medication will be discontinued and patients will receive standard treatment according to the cause of their bleeding. These patients will be followed up for safety only.

*Note: There is no provision in this study to have an expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Female or male cirrhotic patient aged 18 to 75 years.
* Hematemesis and/or melena (suspected to be caused by portal hypertension)
* Time interval <=24 hours between onset of initial hemorrhage and initiation of study drug infusion.
* Time interval <=6 hours between admission and initiation of study drug infusion.
* Anticipated time interval<=12 hours between admission and end of therapeutic endoscopy.
* Unequivocal history of cirrhosis, either documented by at least one of classical clinical signs (abdominal collateral venous circulation, firm liver with a sharp lower liver edge, presence of spider naevi, and/or ascites), or by biochemical and/or Doppler-US signs.
* Written informed consent obtained by the patient or his/her relative(s)

Exclusion Criteria:

* Patient previously included in this study for a prior bleeding episode.
* Patients treated with a vasoactive drug such as octreotide, vasopressin or its analogue for the current episode of bleeding.
* Hepatic encephalopathy Grade IV.
* Balloon tamponade already positioned at admission.
* Known Child-Pugh score >=13
* Pregnant or breast-feeding women.
* Known diffuse hepatocellular carcinoma.
* Known complete portal venous thrombosis.
* Bleeding from esophageal varices within the previous 6 weeks.
* Patient currently enrolled in another therapeutic study, and/or who participated in another clinical study, within the previous 6 weeks.
* Known allergy to somatostatin or somatostatin analogues.
* Previous porto-systemic shunt (TIPS) or orthotopic liver transplantation.
* Patient with known cancer.
* Patient with known chronic renal failure (serum creatinine > 1.5 mg/dl).
* Severe concomitant disease judged by the Investigator as being incompatible with evaluation of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of the early administration of Sanvar® (vapreotide) in association with endoscopic treatment for the control of bleeding at 5 days, i.e. control of initial bleeding and prevention of early re-bleeding, plus survival. | 5 days

SECONDARY OUTCOMES:
To assess the following:
The effect of drug administration before endoscopy assessed by the endoscopic facilitation and control of bleeding at endoscopy, | Endoscopy
Control of bleeding 6 hours after infusion of the study drug (= Tinf + 6h), | Tinf + 6h
Control of bleeding by time periods (Tendo+6h, Tendo+48h and Tendo+ 120h) by Child Pugh class, | Tendo+6h, Tendo+48h and Tendo+ 120h
Number of blood units administered during the 5 days of drug infusion, | 5 days
Safety of treatment | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lim, M.D., Study Chair — Yale University; Tarek Hassanein, M.D., Principal Investigator — University of California, San Diego; Michael B. Fallon, M.D., Principal Investigator — UAB Liver Center, Division of Gastroenterology & Hepatology; Daniel R. Ganger, M.D., Principal Investigator — Northwestern Memorial Hospital; Naga P. Chalasani, M.D., Principal Investigator — Indiana University School of Medicine; Adrian Reuben, M.D., Principal Investigator — Medical University of South Carolina; Paul J. Thuluvath, M.D., Principal Investigator — The Johns Hopkins Hospital & School of Medicine; James F. Trotter, M.D., Principal Investigator — University of Colorado, Denver; Hugo Vargas, M.D., Principal Investigator — Mayo Clinic Scottsdale, Arizona; Samuel Sigal, M.D., Principal Investigator — Weill Medical College of Cornell University; Michele D. Bishop, M.D., Principal Investigator — Mayo Clinic Jacksonville Florida; Gary A. Abrams, M.D., Principal Investigator — Alabama Liver & Digestive Specialists Research Center - Montgomery, AB; Robert S. McFadden, M.D., Principal Investigator — CHRISTUS Santa Rosa Medical Center - San Antonio, TX; Nezam H. Afdhal, M.D., Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA; Jeffrey S. Crippin, M.D., Principal Investigator — Washington University School of Medicine; Alvaro Koch, M.D., Principal Investigator — University of Kentucky Medical Center - Lexington, KY; Kimberly Beavers, M.D., M. Ph., Principal Investigator — Mission Hospitals, Inc. - Asheville, NC; Arun J. Sanyal, M.D., Principal Investigator — Virginia Commonwealth University
Locations (19):
- United States (19):
  - UAB Liver Center, Birmingham, Alabama
  - Alabama Liver & Digestive Specialists, Montgomery, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of California at San Diego, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University, The Feinberg School of Medicine, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins Hospital & School of Medicine, Div. of Gastroenterology & Hepatology, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mission Hospitals, Inc., Asheville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CHRISTUS Santa Rosa Medical Center, San Antonio, Texas
  - Virginia Commonwealth University MCV Campus West Hospital, Richmond, Virginia

REFERENCES:
- [Background] Cales P, Masliah C, Bernard B, Garnier PP, Silvain C, Szostak-Talbodec N, Bronowicki JP, Ribard D, Botta-Fridlund D, Hillon P, Besseghir K, Lebrec D; French Club for the Study of Portal Hypertension. Early administration of vapreotide for variceal bleeding in patients with cirrhosis. N Engl J Med. 2001 Jan 4;344(1):23-8. doi: 10.1056/NEJM200101043440104. PMID 11136956
- See also: N Engl J Med. 2001 Jan 4;344(1):23-8 — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=11136956&query_hl=1&itool=pubmed_docsum